CLINICAL TRIAL: NCT01061216
Title: A Mono-center, Open Label, Randomised 2-period Crossover Study to Compare the Pharmacokinetics and Pharmacodynamics of Continuous Insulin Infusion Administered Either Intradermally or Subcutaneously in Subjects With Type 1 Diabetes Mellitus
Brief Title: Pharmacokinetics/Dynamics of Basal (Continuous) Insulin Infusion Administered Either Intradermally or Subcutaneously
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Becton, Dickinson and Company (Industry)
Responsible Party: Kevin Judge / VP / Corporate Clinical Development and Clinical Operations, Becton Dickinson
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: BDT-09-ADC003; 2009-016164-36 (EudraCT Number)
Record Dates: First submitted 2010-01-29; First posted 2010-02-03 (Estimated); Last update posted 2010-03-10 (Estimated); Status verified 2010-03

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
Keywords: Diabetes; Insulin Therapy; Blood Glucose; Basal insulin; Diabetics
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intradermal insulin infusion (ID) (Experimental)
  Interventions: Device: Intradermal insulin delivery: BD Research Catheter Set
- Subcutaneous insulin infusion (SC) (Active Comparator)
  Interventions: Device: Subcutaneous insulin delivery:ACCU-CHEK Rapid-D Infusion Set

INTERVENTIONS:
Device: Intradermal insulin delivery: BD Research Catheter Set — 1 unit/hr rapid acting insulin delivered intradermally for 6 hours 4 hour washout period (no insulin delivered) 2 units/hr rapid acting insulin delivered intradermally for 6 hours 4 hour washout period (no insulin delivered)
  Arms: Intradermal insulin infusion (ID)
Device: Subcutaneous insulin delivery:ACCU-CHEK Rapid-D Infusion Set — 1 unit per hour of rapid acting insulin infusion for 6 hours 4 hour washout (no insulin delivered) 2 unit per hour of rapid acting insulin infusion for 6 hours 4 hour washout (no insulin delivered)
  Other Names: ACCU-CHEK; Rapid-D Infusion Set (Disetronic, USA)
  Arms: Subcutaneous insulin infusion (SC)

SUMMARY:
The primary objective of this study will be to assess the PK/PD responsiveness of basal ID administered insulin compared to SC, and to determine the safety and local tolerability of extended (two six-hour periods) microneedle insulin delivery (MID) infusion. The primary endpoint will be the PK response to changes in rapid-acting insulin basal infusion rate.

Faster PK transitions coupled with faster PD responsiveness could provide clinical benefit, compared to current subcutaneous insulin infusion. In addition, for nocturnal basal pumping, more rapid insulin offset could decrease the occurrence rate and severity of hypoglycemic episodes.

DETAILED DESCRIPTION:
Twenty (20) male T1 diabetic subjects will be studied under manual partial glucose clamp conditions over a 16 hour infusion period (approximately 36 hours of overall time in clinic). Subjects will be admitted to the clinic the night before their study visit for overnight stabilization in which, via insulin and/or glucose infusions, blood glucose will be stabilized to approximately 140 mg/dL. Subjects will receive as background IV Humulin insulin with an initial dose equivalent to one-half of their usual daily basal insulin dose. In the morning the subjects will start the experimental intervention and have administered a low rate stair-stepped Lispro insulin infusion profile via an infusion pump (Harvard Syringe Pump, Harvard Apparatus).

The profile is designed to examine the initial "on" rate for microneedle insulin delivery, the transition time between basal rate changes and the "off-rate" after insulin cessation. Subjects will receive the same profile by SC infusion on a second clinic day in a randomized order. PK endpoints will be established using timed blood samples. Safety and tolerability at the local infusion site will also be recorded.

In parallel, using a commercially available insulin pump (One Touch "Ping" Insulin Pump, Animas) and an infusion set (either the RCS or a commercially available SC insulin infusion set); a second infusion of insulin diluent will be used to assess the feasibility of longer-term ID infusions (16 hours) as compared to SC.

During each infusion the pumps will control the fluid delivery rate and volume. In addition an in-line pressure transducer will record the pressure and transfer the information to a laptop computer.

Primary Objective:

* To define the PK profile of initiation, rate change, and discontinuation of continuously infused basal insulin administered either intradermally or subcutaneously over two separate infusion periods.

Secondary Objectives:

* Determine the PD effect of the infused insulin as measured by time to glucose rebound following discontinuation of test insulin infusion.
* Assess the safety and tolerability of intradermally infused insulin over two six-hour periods.
* Assess the feasibility of the research catheter set (RCS) for longer-term ID infusion

ELIGIBILITY:
20 Male Type 1 Diabetic Mellitus subjects on Continuous Subcutaneous Insulin Infusion (CSII) therapy.

Inclusion Criteria:

* Understood and signed informed consent obtained before any trial-related activities (trial-related activities are any procedures that would not have been performed during normal management of the subject)
* Type 1 Diabetes mellitus, according to clinical judgment / ADA / WHO-definition (Diabetes Care 2003; 26: 5-20) for at least 1 year
* Current treatment:Insulin Pump
* Age in the range of greater than or equal to 18 and less than or equal to 55 years
* Body mass index (BMI) less than or equal to 32 kg/m²
* HbA1c less than or equal to 9.0 %
* Able and willing to adhere to the study procedures for the entire trial period
* Negative test results for hepatitis C antibodies, hepatitis B surface antigen and HIV at screening.

Exclusion Criteria:

* Previous participation in this trial or participation in a clinical trial within 3 months prior screening examination
* Any symptoms suggestive of, or a diagnosis or treatment for gastroparesis
* Abnormalities in renal function (e.g. serum creatinine >1.2 mg/dl) or judged by the investigator that would pose a problem of clearance of injected insulin
* Proliferative retinopathy or maculopathy that has required acute treatment within the last six months
* Acute and severe illness apart from diabetes mellitus as judged by the investigator
* Abnormalities in the laboratory parameters if judged as clinically significant by the investigator. In particular, subjects with GOT/GPT >3x, thrombocyte count <100/nL, INR >1.3, PTT >50 sec. will not be permitted to enter the study.
* Clinically significant abnormalities in the ECG
* Recurrent major hypoglycemia or hypoglycemic unawareness as judged by the investigator
* Lipodystrophy which in the judgment of the investigator would pose a problem in terms of variability of absorption of injected insulin
* Use of systemic corticoids for the last three months prior to screening examination or treatment with medication known to interfere with glucose metabolism such as non-selective ß-blockers, or mono amine oxidase (MAO) inhibitors, ACE-inhibitors or thiazides, unless medical treatment having existed for at least three month prior screening examination
* Any disease requiring use of anti-coagulants
* Impaired hepatic or renal functions as judged by the investigator
* Cardiac problems as judged by the investigator
* Uncontrolled hypertension (treated or untreated) as judged by the investigator (RRsyst. >140 mmHg, RRdiast. > 90 mmHg)
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or co-operation
* Current addiction to alcohol or substances of abuse as determined by the investigator
* Allergy to plaster/adhesive
* Any other condition that the investigator feels would interfere with trial participation or evaluation of results.
* Donation of any blood or plasma in the past month or in excess of 500 mL within the 12 weeks preceding screening
* Subjects with a history of deep leg vein thrombosis or with frequent appearance of deep leg vein thrombosis in 1st degree relatives as judged by the investigator

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Insulin measurements will be used to compute PK model parameters: absorption rate(s) and elimination rate using an appropriate transport model. | 20 hours

SECONDARY OUTCOMES:
Pharmacodynamic glycemic parameters will be as follows: time from insulin infusion onset to glycemic nadir; time from test insulin shutoff to return to baseline glucose; amount of additional drop in blood glucose following test insulin infusion shutoff | 20 hours
Evidence of safety and tolerability of intradermally infused insulin | 26 hours
Feasibility of RCS for longer-term ID infusion | 16 hours

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Kapitza, Dr. med., Principal Investigator — Profil Institut für Stoffwechselforschung GmbH
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, Germany